CLINICAL TRIAL: NCT05857826
Title: Effects of Soft Tissue Release With and Without Vaginal Dilators on Pain and Sexual Function in Women With Genito Pelvic Pain
Brief Title: Soft Tissue Release With and Without Vaginal Dilators on Pain and Sexual Function in Genitio Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0526
Record Dates: First submitted 2023-04-18; First posted 2023-05-15 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Genito-Pelvic Pain/Penetration Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- soft tissue release with vaginal dilators (Experimental): Group A will receive soft tissue release with vaginal diltors. Soft tissue release consists of myofacial release and deep intervaginal massage.Triggers points can be released vaginally or rectally they are so painfyul on palpation deep massage of pelvic floor muscle
  Interventions: Other: soft tissue release; Other: vaginal dilators
- soft tissue release only (Active Comparator): will receive only soft tissue release using trigger point release vaginally or rectally and deep intervaginal massage
  Interventions: Other: soft tissue release

INTERVENTIONS:
Other: soft tissue release — Patient will be asked to lie in hook lying position using a clean glove will apply some water based lubricant gently sweep vaginal muscle from superficial to deep until find a trigger point press it and release it using circle motion for 1 to 2 minute until the trigger point is completely released.
Other: vaginal dilators — Vaginal dilators will be used according to the patient's condition starting from small sizes to the wider ones.
  Arms: soft tissue release with vaginal dilators

SUMMARY:
Study will be a randomized clinical trial which will incorporate two different interventions soft tissue release and vaginal dilators use would be administered to the women with genito pelvic pain. Subjects meeting the predetermined inclusion criteria will be divided into two groups using lottery method. Assessment will be done using GPPPD, Vancouver Visual Analogue Scale, female sexual function index and pelvic floor impact questionnaire. Subjects in one group will be treated with soft tissue release and vaginal dilators. And the other will be treated with soft tissue release only. Each subject will receive a total 09 treatment sessions, with 03 treatment sessions per week. Measurements will be recorded at baseline, 5th and 9th treatment session.

DETAILED DESCRIPTION:
Painful sexual intercourse is a common female health problem. It is a complex disorder that often goes neglected. It can be further categorized into superficial or deep, and primary or secondary. Superficial is limited to the vulva or vaginal entrance, while deep means the extension of pain into the deeper parts of the vagina or lower pelvis. Deep dyspareunia is frequently associated with deep penetration. Primary pain initiates at the start of sexual intercourse, while in secondary, pain begins after some time of pain free sexual activity This study will be a randomized clinical trial which will incorporate two different interventions soft tissue release and vaginal dilators use would be administered to the women with genito pelvic pain. Subjects meeting the predetermined inclusion criteria will be divided into two groups using lottery method. Assessment will be done using GPPPD, Vancouver Visual Analogue Scale, female sexual function index and pelvic floor impact questionnaire . Subjects in one group will be treated with soft tissue release and vaginal dilators. And the other will be treated with soft tissue release only. Each subject will receive a total 09 treatment sessions, with 03 treatment sessions per week. Measurements will be recorded at baseline, 5th and 9th treatment session. Recorded values will be analyzed for any change using SPSS21.

ELIGIBILITY:
Inclusion Criteria:

* Women age 20 to 40 years
* Patient fulfilling DSM5 GPPPD criteria
* Pain in genitals before during or after intercourse
* Pain greater than 4 on a 10cm visual analogue scale

Exclusion Criteria:

* • History of pathological conditions like infections

  * Endometriosis
  * Tumors
  * Major psychiatric disorders
  * Painful bladder syndrome
  * Surgery of pelvic organs
  * Any ongoing treatment of genito pelvic pain.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Female sexual function index | up to 3 weeks
  The Female Sexual Function Index (FSFI) is a very well-worded sexual function screen with excellent psychometric qualities. However, some aspects of the scoring procedures pose conceptual and statistical problems, which we illustrate in part by way of an empirical example. The recommended solutions should further strengthen the utility and validity of this instrument
Visual analogue scale | up to 3 weeks
  Describes the construction of visual analogue scale that could be used with critically ill patients, the structural and visual cues on this VAS allow for exact placement of the template and reliable measurements. Rates pain from 1 to 10.
Pelvic floor impact questionnaire | up to 3 weeks
  The Pelvic Floor Distress Inventory-20 and Pelvic Floor Impact Questionnaire-7 are valid, reliable, and responsive short forms of 2 condition-specific quality-of-life questionnaires for women with pelvic floor disorders

CONTACTS AND LOCATIONS:
Overall Officials: Asma Ambreen, MS*, Principal Investigator — Riphah International University
Locations (1):
- Lahore general hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Trahan J, Leger E, Allen M, Koebele R, Yoffe MB, Simon C, Alappattu M, Figuers C. The Efficacy of Manual Therapy for Treatment of Dyspareunia in Females: A Systematic Review. J Womens Health Phys Therap. 2019 Jan-Mar;43(1):28-35. doi: 10.1097/jwh.0000000000000117. PMID 34135723
- [Background] Fisher KA. Management of dyspareunia and associated levator ani muscle overactivity. Phys Ther. 2007 Jul;87(7):935-41. doi: 10.2522/ptj.20060168. Epub 2007 May 1. PMID 17472951
- [Background] Antosh DD, Gutman RE, Park AJ, Sokol AI, Peterson JL, Kingsberg SA, Iglesia CB. Vaginal dilators for prevention of dyspareunia after prolapse surgery: a randomized controlled trial. Obstet Gynecol. 2013 Jun;121(6):1273-1280. doi: 10.1097/AOG.0b013e3182932ce2. PMID 23812462
- [Background] Rosenbaum TY. Physiotherapy treatment of sexual pain disorders. J Sex Marital Ther. 2005 Jul-Sep;31(4):329-40. doi: 10.1080/00926230590950235. PMID 16020150
- [Background] Both S, Brauer M, Weijenborg P, Laan E. Effects of Aversive Classical Conditioning on Sexual Response in Women With Dyspareunia and Sexually Functional Controls. J Sex Med. 2017 May;14(5):687-701. doi: 10.1016/j.jsxm.2017.03.244. Epub 2017 Mar 31. PMID 28372937
- [Background] Ghaderi F, Bastani P, Hajebrahimi S, Jafarabadi MA, Berghmans B. Pelvic floor rehabilitation in the treatment of women with dyspareunia: a randomized controlled clinical trial. Int Urogynecol J. 2019 Nov;30(11):1849-1855. doi: 10.1007/s00192-019-04019-3. Epub 2019 Jul 8. PMID 31286158
- [Background] Meyer-Bahlburg HF, Dolezal C. The female sexual function index: a methodological critique and suggestions for improvement. J Sex Marital Ther. 2007 May-Jun;33(3):217-24. doi: 10.1080/00926230701267852. PMID 17454519
- [Background] Cline ME, Herman J, Shaw ER, Morton RD. Standardization of the visual analogue scale. Nurs Res. 1992 Nov-Dec;41(6):378-80. No abstract available. PMID 1437591